CLINICAL TRIAL: NCT02847182
Title: Efficacy of Intravenous Umbilical Cord Blood Infusion as Cell Therapy for Children With Autism Spectrum Disorder (ASD): Duke ACT
Brief Title: Cord Blood Infusion for Children With Autism Spectrum Disorder
Acronym: Duke ACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Chief Scientific Officer, Robertson Clinical and Translational Cell Therapy Program; Director, Pediatric Blood and Marrow Transplant Program and Carolinas Cord Blood Bank, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00070514
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Autism Spectrum Disorder; ASD; Autism; PDD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cord Blood Infusion (best source) (Experimental): Subjects will be randomized to receive a cord blood infusion at the baseline or 6 month visit. The cord blood will be autologous (if available) or unrelated cord blood.
  Interventions: Biological: Cord Blood Infusion; Biological: Placebo
- Placebo Infusion (Placebo Comparator): Subjects will be randomized to receive a placebo infusion at the baseline or 6 month visit. The placebo is an acellular media product similar in both appearance and odor.
  Interventions: Biological: Cord Blood Infusion; Biological: Placebo

INTERVENTIONS:
Biological: Cord Blood Infusion
Biological: Placebo

SUMMARY:
This is a single site, prospective, randomized, double-blind study of a single intravenous autologous or allogeneic, unrelated cord blood (CB) infusion in children ages 2-7 years with Autism Spectrum Disorder (ASD). Participants will be randomly assigned to Sequence A, consisting of a single infusion of CB cells at baseline followed 6 months later by a single infusion of placebo, or Sequence B, consisting of an infusion of placebo at baseline followed 6 months later by an infusion of CB cells. All participants will ultimately be treated with CB cells at some point during the study. Participants with an available qualified autologous CB unit will receive autologous cells, and those without a suitable autologous CB unit available will receive cells from a ≥4/6 HLA-matched, ABO-matched allogeneic, unrelated donor CB unit from the Carolinas Cord Blood Bank. All infusions will be double-blinded. The primary outcomes will be assessed 6 months after the initial infusion in the sequence. Additional testing for secondary exploratory analyses will be performed at 12 months. Duration of study participation will be 12 months from the time of baseline infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years to ≤ 7 years (7 years, 364 days) at the time of visit 1
2. Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using the DSM-5 Checklist
3. Fragile X testing performed and negative
4. Available and qualified umbilical cord blood unit with a minimum banked total nucleated cell dose of ≥ 2.5 x 107 cells/kg that meets criteria outlined in Section 6.0, either:

   * Autologous umbilical cord blood unit OR
   * ≥4/6 HLA-matched and ABO/Rh-matched allogeneic unrelated umbilical cord blood unit from the Carolinas Cord Blood Bank
5. Stable on current psychiatric medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product
6. Normal absolute lymphocyte count (≥1500/uL)
7. Participant and parent/guardian are English speaking
8. Able to travel to Duke University two times (baseline and 6 months post-baseline), and parent/guardian is able to participate in interim surveys and interviews
9. Parental consent

Exclusion Criteria:

1. General:

   * Review of medical records indicates ASD diagnosis not likely
   * Known diagnosis of any of the following coexisting psychiatric conditions: depression, bipolar disorder, schizophrenia, obsessive compulsive disorder, Tourette syndrome
   * Screening data suggests that participant would not be able to comply with the requirements of the study procedures, including study outcome measures, as assessed by the study team
   * Family is unwilling or unable to commit to participation in all study-related assessments, including follow up for approximately 12 months
   * Sibling is enrolled in this (DukeACT) study
2. Genetic:

   * Records indicate that child has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy b. Known pathogenic copy number variation (CNV) associated with ASD (e.g., 16p11.2, 15q13.2, 2q13.3)
3. Infectious:

   * Known active central nervous system infection
   * Evidence of uncontrolled infection based on records or clinical assessment
   * HIV positivity
4. Medical:

   * Known metabolic disorder
   * Known mitochondrial dysfunction
   * History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome, or other similar chronic seizure disorder
   * Active malignancy or prior malignancy that was treated with chemotherapy
   * History of a primary immunodeficiency disorder
   * History of autoimmune cytopenias (i.e., ITP, AIHA)
   * Coexisting medical condition that would place the child at increased risk for complications of sedation or other study procedures
   * Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
   * Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
   * Impaired renal or liver function as determined by serum creatinine >1.5mg/dL or total bilirubin >1.3mg/dL, except in patients with known Gilbert's disease
   * Significant hematologic abnormalities defined as: Hemoglobin <10.0 g/dL, White blood count < 3,000 cells/mL, absolute lymphocyte count <1000/uL, Platelets <150 x 10e9/uL
   * Evidence of clinically relevant physical dysmorphology indicative of a genetic syndrome as assessed by the PIs or other investigators, including a medical geneticist or psychiatrists trained in identifying dysmorphic features associated with neurodevelopmental conditions
5. Current/Prior Therapy:

   * History of prior cell therapy
   * Current or prior use of immune globulins or other anti-inflammatory medications with the exception of non steroidal anti-inflammatory medications
   * Current or prior immunosuppressive therapy
   * No systemic steroid therapy that has lasted >2 weeks, and no systemic steroids within 3 months prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke Medicine
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Simhal AK, Carpenter KLH, Kurtzberg J, Song A, Tannenbaum A, Zhang L, Sapiro G, Dawson G. Changes in the geometry and robustness of diffusion tensor imaging networks: Secondary analysis from a randomized controlled trial of young autistic children receiving an umbilical cord blood infusion. Front Psychiatry. 2022 Oct 20;13:1026279. doi: 10.3389/fpsyt.2022.1026279. eCollection 2022. PMID 36353577

RESULTS

PARTICIPANT FLOW:
Groups:
- Cord Blood Infusion, Then Placebo Infusion: Subjects will be randomized to receive a cord blood infusion at the baseline visit, followed by a placebo infusion at 6 months. The cord blood will be autologous (if available) or unrelated cord blood. The placebo is an acellular media product similar in both appearance and odor.
  Cord Blood Infusion
  Placebo
- Placebo Infusion, Then Cord Blood Infusion: Subjects will be randomized to receive a placebo infusion at the baseline visit, followed by a cord blood infusion at 6 months. The placebo is an acellular media product similar in both appearance and odor. The cord blood will be autologous (if available) or unrelated cord blood.
  Cord Blood Infusion
  Placebo
Period: Overall Study
Arm/Group | Cord Blood Infusion, Then Placebo Infusion | Placebo Infusion, Then Cord Blood Infusion
Started | 119 | 61
First Intervention (6 Months) | 119 | 61
Second Intervention (6 Months) | 61 | 119
Completed | 119 | 60
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The protocol-specified pilot subjects, both randomized to placebo, were also mistakenly enrolled several days after their 8th birthday, in violation of the age-related inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cord Blood Infusion, Then Placebo Infusion | Placebo Infusion, Then Cord Blood Infusion | Total
Number analyzed (Participants) | 119 | 61 | 180
Age, Continuous [Median (Full Range); unit: years] | 5.30 [2.39 to 8.00] | 5.24 [2.31 to 8.13] | 5.29 [2.31 to 8.13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 98 | 45 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 6 | 32
  Not Hispanic or Latino | 93 | 55 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-White | 24 | 17 | 41
  White | 95 | 44 | 139
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 119 | 61 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Communication as Measured by the Vineland Adaptive Behavior Scales, Third Edition (VABS-3)
Description: The Vineland Adaptive Behavior Scales, Third Edition (VABS-3) Socialization domain standard score has mean=100 and standard deviation=15 (range: 20-140). Higher scores indicate better developed adaptive social behavior. The change in the Socialization domain standard score was calculated for each participant from Baseline to Month 6. Changes in the Socialization standard score are indicative of skill acquisition relative to chronologically aged peers of the same sex. Thus, a zero (no change) represents change consistent with what is expected. An increase represents acquisition of more skills over time than would be expected. Participants who experience a decrease in Socialization standard score may still have acquired skills although not at the rate expected based on their age and sex.
Time Frame: Baseline, 6 months
Population: Four subjects randomized to placebo were not included in the efficacy analyses. Two were pre-specified exclusions (defined as pilot subjects in the protocol) and two were found ineligible after enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cord Blood Infusion - 6 Months: Subjects will be randomized to receive a cord blood infusion at the baseline visit. The cord blood will be autologous (if available) or unrelated cord blood.
  Cord Blood Infusion
- Placebo Infusion - 6 Months: Subjects will be randomized to receive a placebo infusion at the baseline visit. The placebo is an acellular media product similar in both appearance and odor.
  Placebo
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale | 3.13 (8.76) | 1.98 (8.41)
Statistical Analysis 1: Comparison: Cord Blood Infusion - 6 Months vs Placebo Infusion - 6 Months; Null hypothesis: The mean of the 6-month change in VABS-II Socialization Subscale Standard Score is the same for the Cord Blood and Placebo groups; Test type: Superiority; p = 0.83, t-test, 2 sided; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-1.58 to 3.86]

2. Secondary Outcome: Change in Vineland Socialization Domain Raw Score
Description: There are 3 raw scores within the Socialization domain of the VABS-3. These are the Interpersonal Relationships Raw Score (range: 0-86), the Play and Leisure Raw Score (range: 0-72), and the Coping Skills Raw Score (range: 0-66). Higher numbers on all three scores reflect better functioning in each area. Each raw score is the sum of the item scores in the respective subdomain of Socialization skills. The items are scored as follows: 2=usually present, 1=sometimes present, 0= never present. The item scores are assigned by a trained interviewer who interviews the parent of the child participating in the study. The change in raw score was calculated for each participant from Baseline to Month 6. Positive scores indicate improvement over time whereas negative scores indicate worsening, and zero indicates no change. The scores are not norm-referenced.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale
  Interpersonal Relationships Raw Score | 5.40 (9.13) | 4.11 (9.42)
  Play and Leisure Raw Score | 4.76 (9.84) | 3.09 (7.68)
  Coping Skills Raw Score | 3.82 (7.54) | 2.91 (7.21)

3. Secondary Outcome: Change in Vineland Socialization Domain Age Equivalent
Description: There are 3 age equivalent scores within the Socialization domain of the VABS-3: the Interpersonal Relationships Age Equivalent, the Play and Leisure Age Equivalent, and the Coping Sills Age Equivalent. An individual participant's age equivalent represents the chronological age (in years:months) at which their score would be considered normative. The age equivalent ranges are 0:0-22:0, 0:0-20:0, and 2:0-22:0 for the Interpersonal Relationships, Play and Leisure and Coping Skills age equivalents, respectively. The change in this age equivalent was calculated for each participant from Baseline to Month 6 and expressed as a number of months. Positive scores indicate increases in the age equivalent of the participant's social communication skills over time and are considered an improvement. Negative scores indicate decreases in the age equivalent of the participant's social communication skills and are considered worsening, and zero indicates no change.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
months
  Interpersonal Relationships Age Equivalent Score | 0.37 (0.72) | 0.19 (0.79)
  Play and Leisure Age Equivalent Score | 0.41 (1.17) | 0.30 (1.21)
  Coping Skills Age Equivalent Score | 0.26 (0.77) | 0.18 (0.89)

4. Secondary Outcome: Change in Pervasive Developmental Disorder Behavior Inventory (PDD-BI) Composite Standard Score (Parent Questionnaire)
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The PDD-BI assesses both social impairments and development of pro-social skills that are integral to improved reciprocal social behavior. The PDD-BI renders T scores (mean=50, standard deviation=10) based on comparisons to a standardized ASD population. The Autism Composite T score ranges from 10-100. The typical child with autism scores between 40-60.Higher scores indicate more severe autism symptoms and lower scores reflect milder symptoms. Change in this score from Baseline to Month 6 was calculated for each participant. Negative change scores indicate improvement in autism symptoms over time whereas positive scores indicate worsening of symptoms, and zero indicates no change in symptoms.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale | -6.65 (10.44) | -6.12 (8.82)

5. Secondary Outcome: Change in Clinical Global Impressions - Severity of Illness (CGI-S) Score, Clinician Assessment
Description: The CGI-S is a 7 point scale completed at the baseline and 6-month visits that requires the clinician to rate the severity of the participant's symptoms of autism at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. There are 3 CGI-S scores: the Social Communication Score, the Restricted and Repetitive Behaviors Score, and the Overall Score. The clinician's rates the severity of autism symptoms - 1, normal, no symptoms; 2, borderline level of symptoms; 3, mild symptoms; 4, moderate symptoms; 5, marked symptoms; 6, severe symptoms; or 7, extremely severe symptoms. Increases in the change score represent increases in symptom severity, decreases in the change score indicate improvement, and zero indicates no change.
Time Frame: Baseline, 6 months
Population: Four subjects randomized to placebo were not included in the efficacy analyses. Two were pre-specified exclusions (defined as pilot subjects in the protocol) and two were found ineligible after enrollment. Two additional subjects were excluded from the Cord Blood group because they were missing assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 117 | 57
score on a scale
  Social Communication Score | -0.11 (0.58) | -0.19 (0.52)
  Restricted, Repetitive Behaviors Score | -0.25 (0.73) | -0.18 (0.73)
  Overall Score | -0.15 (0.57) | -0.26 (0.58)

6. Secondary Outcome: Clinical Global Impressions - Global Improvement (CGI-I) Score, Clinician Assessment
Description: The CGI-I is a 7 point scale that requires the clinician to assess how much the participant's autism symptoms have improved or worsened relative to a baseline assessment. The symptoms are rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. There are three separate CGI-I ratings: social communicative functioning, restricted/repetitive interests and behaviors, and overall improvement.
Time Frame: Baseline, 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 117 | 57
Participants
  Social Communicative Functioning: 1=Very Much Improved | 0 | 0
  Social Communicative Functioning: 2=Much Improved | 26 | 9
  Social Communicative Functioning: 3=Minimally Improved | 30 | 16
  Social Communicative Functioning: 4=No Change | 58 | 31
  Social Communicative Functioning: 5=Minimally Worse | 3 | 1
  Social Communicative Functioning: 6=Much Worse | 0 | 0
  Restricted/repetitive Interests and Behaviors: 1=Very Much Improved | 1 | 0
  Restricted/repetitive Interests and Behaviors: 2=Much Improved | 17 | 11
  Restricted/repetitive Interests and Behaviors: 3=Minimally Improved | 29 | 10
  Restricted/repetitive Interests and Behaviors: 4=No Change | 59 | 29
  Restricted/repetitive Interests and Behaviors: 5=Minimally Worse | 10 | 7
  Restricted/repetitive Interests and Behaviors: 6=Much Worse | 1 | 0
  Overall Score: 1=Very Much Improved | 1 | 0
  Overall Score: 2=Much Improved | 26 | 11
  Overall Score: 3=Minimally Improved | 37 | 18
  Overall Score: 4=No Change | 47 | 27
  Overall Score: 5=Minimally Worse | 6 | 1
  Overall Score: 6=Much Worse | 0 | 0

7. Secondary Outcome: Change in Expressive One-Word Picture Vocabulary Test (Clinician Assessment)
Description: This Expressive One-Word Picture Vocabulary Test is a standardized evaluation of the child's expressive one-word vocabulary by a trained clinician. It tests an individual's ability to name, with one word, objects, actions, and concepts when presented with color illustrations. Higher EOWPVT standard scores reflect a better vocabulary. The minimum score is age-dependent (years:months) as follows. For a child age 2:0 to 2:1 the minimum is 65; age 2:2-2:3 (min=62); age 2:4-2:5 (min=60); age 2:6-2:7 (min=58); age 2:8-2:9 (min=57); age 2:10-2:11 (min=56); age 3:0 and older (min=55). The maximum possible score across all ages is 145. The change in score from Baseline to Month 6 was the outcome measure. Increases reflect increases in vocabulary skills, decreasing reflect decreases in vocabulary skills, and zero reflects no change.
Time Frame: Baseline, 6 months
Population: Four subjects randomized to placebo were not included in the efficacy analyses. Two were pre-specified exclusions (defined as pilot subjects in the protocol) and two were found ineligible after enrollment. Three additional subjects were excluded from the Cord Blood group because they were missing assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 116 | 57
score on a scale | 0.89 (7.48) | 1.88 (10.18)

8. Secondary Outcome: Change in Vineland Adaptive Behavior Scales II (VABS-II) Communication Subscale Standard Score
Description: The VABS-II measures adaptive functioning in socialization, communication, daily living, and motor skills. The Communication subscale standard score is derived by summing norm-referenced (by age group and sex) v-scale scores (mean=15, standard deviation=3) from the Receptive, Expressive, and Written communication subdomains and standardizing this sum to a normal distribution with mean=100 and standard deviation=15. Changes in the Communication standard score are indicative of skill acquisition relative to chronologically aged peers of the same sex. Thus, a zero (no change) represents change consistent with what is expected. An increase represents acquisition of more skills over time than would be expected. Participants who experience a decrease in Communication standard score may still have acquired skills although not at the rate expected based on their age and sex.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale | 2.87 (8.95) | 2.81 (9.68)

9. Secondary Outcome: Change in Vineland Adaptive Behavior Scales II (VABS-II) Daily Living Subscale Standard Score
Description: The VABS-II measures adaptive functioning in socialization, communication, daily living, and motor skills. The Daily Living standard score is derived by summing norm-referenced (by age group and sex) v-scale scores (mean=15, standard deviation=3) from the Personal, Domestic and Community subdomains and standardizing this sum to a normal distribution with mean=100 and standard deviation=15. Changes in the Daily Living standard score are indicative of skill acquisition relative to chronologically aged peers of the same sex. Thus, a zero (no change) represents change consistent with what is expected. An increase represents acquisition of more skills over time than would be expected. Participants who experience a decrease in Daily Living standard score may still have acquired skills although not at the rate expected based on their age and sex.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale | 2.21 (6.89) | 2.49 (7.41)

10. Secondary Outcome: Change in Vineland Adaptive Behavior Scales II (VABS-II) Composite Score
Description: The Vineland Adaptive Behavior Scales II (VABS-II) measures adaptive functioning in socialization, communication, daily living, and motor skills. The Adaptive Behavior Composite provides an overall summary of adaptive behavior across all of the domains. Each participant's score is standardized to a normal distribution with mean=100 and standard deviation=15. Positive scores indicate an increase in the Adaptive Behavior Composite Score over time whereas negative scores indicate decrease in the Adaptive Behavior Composite Score, and zero indicates no change in the Adaptive Behavior Composite Score.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
score on a scale | 2.34 (5.93) | 2.09 (6.05)

11. Secondary Outcome: Change in Pervasive Developmental Disorder Behavior Inventory (PDD-BI) Repetitive, Ritualistic and Pragmatic Problems T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Repetitive, Ritualistic and Pragmatic Problems T-Score (mean=50, standard deviation=10) measures a broad range of behavioral problems associated with autism. The score ranges from 26-100 in patients aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -5.50 (10.38) | -5.18 (8.47)

12. Secondary Outcome: Change in PDD-BI Approach/Withdrawal Problems T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Approach/Withdrawal Problems T-Score (mean=50, standard deviation=10) measures a broad range of behavioral problems associated with autism. The score ranges from 27-100 in patients aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -5.42 (10.60) | -4.86 (8.09)

13. Secondary Outcome: Change in PDD-BI Sensory/Perceptual Approach Behaviors T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Sensory/Perceptual Approach Behaviors T-score (mean=50, standard deviation=10) includes behaviors that are largely non-communicative and involve approach toward asocial stimuli. The score ranges from 31 to 86 in patients aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -4.13 (6.80) | -2.75 (6.66)

14. Secondary Outcome: Change in PDD-BI Ritualisms/Resistance to Change T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Ritualisms/Resistance to Change T-Score (mean=50, standard deviation=10) describes behaviors that communicate the child's desires to carry out rituals or to communicate dissatisfaction with a change in the environment or routine. The score ranges from 34 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -5.66 (7.62) | -5.00 (8.61)

15. Secondary Outcome: Change in PDD-BI Social Pragmatic Problems T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Social Pragmatic Problems T-Score (mean=50, standard deviation=10) measures the difficulties children with autism have in either reacting to the approaches of others, understanding social conventions, or initiating social interactions with others. The score ranges from 29 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -3.66 (11.36) | -3.33 (8.78)

16. Secondary Outcome: Change in PDD-BI Semantic/Pragmatic Problems T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Semantic/Pragmatic Problems T-Score (mean=50, standard deviation=10) assesses the difficulties children with autism have in using spoken language to indicate comprehension, communicate meaning, respond to the interests of others, and sustain a conversation. The score ranges from 34 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -3.82 (7.51) | -3.68 (7.90)

17. Secondary Outcome: Change in PDD-BI Arousal Regulation Problems T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Arousal Regulation Problems T-Score (mean=50, standard deviation=10) measures behaviors that are largely non-communicative or unresponsive and reflect emotional constriction, the apparent seeking of kinesthetic sensation, and, in the parent version, difficulty with sleep regulation. The score ranges from 26 to 77 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -4.34 (7.49) | -5.02 (7.28)

18. Secondary Outcome: Change in PDD-BI Specific Fears T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Specific Fears T-Score (mean=50, standard deviation=10) measures behaviors that communicate the fears and anxieties associated with withdrawal from social or asocial stimuli. The score ranges from 36 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -4.24 (8.81) | -3.00 (8.82)

19. Secondary Outcome: Change in PDD-BI Aggressiveness T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Aggressiveness T-Score (mean=50, standard deviation=10) assesses the aggressive approach toward self or others, as well as the negative mood changes that are often associated with such behaviors. The score ranges from 36 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of severity. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect worsening of problem behaviors, decreases indicate improvement, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | -4.31 (11.41) | -1.79 (9.07)

20. Secondary Outcome: Change in PDD-BI Expressive Social Communication Abilities T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Expressive Social Communication Abilities T-Score (mean=50, standard deviation=10) measures a broad range of social communication skills affected by autism. The score ranges from 20 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of competence. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect improvement, decreases indicate worsening, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | 3.20 (5.34) | 2.74 (5.55)

21. Secondary Outcome: Change in PDD-BI Receptive/Expressive Social Communication Ability T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Receptive/Expressive Social Communication Ability T-Score (mean=50, standard deviation=10) measures a broad range of social communication skills affected by autism. The score ranges from 20 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of competence. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect improvement, decreases indicate worsening, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | 2.99 (5.09) | 2.28 (5.16)

22. Secondary Outcome: Change in PDD-BI Social Approach Behaviors T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Social Approach Behaviors T-Score (mean=50, standard deviation=10) assesses those social communication skills that are notoriously difficult for children with autism (e.g., eye contact, joint attention, effective use of gesture, imaginative skills). The score ranges from 14 to 93 for participants aged 2-8 years. Higher values indicate increasing levels of competence. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect improvement, decreases indicate worsening, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | 3.92 (6.46) | 3.23 (5.99)

23. Secondary Outcome: Change in PDD-BI Expressive Language T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Expressive Language T-Score (mean=50, standard deviation=10) assesses the ability of the child to speak the sounds associated with the English language and to use words and sentences that indicate his or her competence with grammar, tone of voice, and the pragmatic aspects of communicating with others. The score ranges from 28 to 100 for participants aged 2-8 years. Higher values indicate increasing levels of competence. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect improvement, decreases indicate worsening, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | 2.03 (4.92) | 1.86 (5.07)

24. Secondary Outcome: Change in PDD-BI Learning, Memory, and Receptive Language T-Score
Description: The PDD-BI is an informant-based rating scale that assesses problem behaviors as well as appropriate social, language, and learning/memory skills. The Learning, Memory, and Receptive Language T-Score (mean=50, standard deviation=10) assesses two areas of variable competence in children with autism: (a) memory and (b) receptive language. The score ranges from 22 to 88 for participants aged 2-8 years. Higher values indicate increasing levels of competence. The change in this score from Baseline to Month 6 was calculated for each participant. Increases in the change score reflect improvement, decreases indicate worsening, and zero indicates no change.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months
Number analyzed (Participants) | 119 | 57
T score | 2.02 (5.45) | 1.05 (5.37)

25. Secondary Outcome: Number of Participants With Infusion Reactions
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Cord Blood Infusion - 12 Months: Subjects will be randomized to receive a cord blood infusion at the baseline visit. The cord blood will be autologous (if available) or unrelated cord blood.
  Cord Blood Infusion
- Placebo Infusion - 12 Months: Subjects will be randomized to receive a placebo infusion at the baseline visit. The placebo is an acellular media product similar in both appearance and odor.
  Placebo
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 61 | 119
Participants | 2 | 1

26. Secondary Outcome: Severity of Infusion Reactions
Description: Grade/severity will be assessed according to CTCAE v4.0 guidelines
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 61 | 119
Participants
  Mild | 2 | 0
  Moderate | 0 | 1
  Severe | 0 | 0

27. Secondary Outcome: Number of Participants With Product-related Infections
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 61 | 119
Participants | 0 | 0

28. Secondary Outcome: Severity of Product-related Infections
Description: Grade/severity will be assessed according to CTCAE v4.0 guidelines
Time Frame: 12 months
Population: There were no product-related infections in the study.
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Evidence of Alloimmunization Via Anti-HLA (Human Leukocyte Antigen) and Anti-RBC (Red Blood Cell) Antibodies and Nonspecific Markers of Systemic Inflammation (ESR, CRP)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 61 | 119
Participants | 0 | 0

30. Secondary Outcome: Incidence of Graft vs. Host Disease
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 61 | 119
Participants | 0 | 0

31. Secondary Outcome: Severity of Graft vs. Host Disease
Description: Grade/severity will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0 guidelines.
Time Frame: 12 months
Population: There were no cases of graft vs. host disease in the study.
Arm/Group | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Incidence of Unexpected Adverse Events, by Relation to Study Product
Time Frame: 6 months,12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 119 | 61 | 61 | 119
Participants
  Related | 0 | 0 | 0 | 0
  Unrelated | 5 | 1 | 0 | 2

33. Secondary Outcome: Severity of Unexpected Adverse Events, by Relation to Study Product
Description: Grade/severity will be assessed according to CTCAE v4.0 guidelines
Time Frame: 6 months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
Number analyzed (Participants) | 119 | 61 | 61 | 119
Participants
  Mild : Related | 0 | 0 | 0 | 0
  Mild : Unrelated | 2 | 0 | 0 | 2
  Moderate : Related | 0 | 0 | 0 | 0
  Moderate : Unrelated | 3 | 1 | 0 | 0
  Severe : Related | 0 | 0 | 0 | 0
  Severe : Unrelated | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months and 12 months
Description: Adverse events collected on Safety Population (all 180 participants). Participants were randomized to receive a single infusion of umbilical cord blood or placebo and evaluated at six months. Participants then received a second infusion in a blinded fashion (placebo for participants initially randomized to cord blood, and cord blood for participants initially randomized to placebo). Participants were then followed for an additional 6 months for safety data collection.
Arm/Group | Cord Blood Infusion - 6 Months | Placebo Infusion - 6 Months | Cord Blood Infusion - 12 Months | Placebo Infusion - 12 Months
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/61 | 0/61 | 0/119
Serious Adverse Events (participants affected / at risk) | 3/119 | 3/61 | 3/61 | 2/119
Other Adverse Events (participants affected / at risk) | 97/119 | 51/61 | 41/61 | 83/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cord Blood Infusion - 6 Months (N=119) | Placebo Infusion - 6 Months (N=61) | Cord Blood Infusion - 12 Months (N=61) | Placebo Infusion - 12 Months (N=119)
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 1 | 0
Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infection (Psychiatric disorders) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cord Blood Infusion - 6 Months (N=119) | Placebo Infusion - 6 Months (N=61) | Cord Blood Infusion - 12 Months (N=61) | Placebo Infusion - 12 Months (N=119)
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Distractibility (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysphemia (Psychiatric disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Adenoidectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Ear tube removal (Surgical and medical procedures) | 0 | 1 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Excessive eye blinking (Eye disorders) | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 3
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 3 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 2
Fatigue (General disorders) | 3 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 2 | 0 | 1
Pyrexia (General disorders) | 11 | 8 | 8 | 5
Thirst (General disorders) | 2 | 0 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 4 | 3 | 1 | 9
Body tinea (Infections and infestations) | 2 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 5 | 1 | 0 | 2
Croup infectious (Infections and infestations) | 1 | 1 | 0 | 2
Ear infection (Infections and infestations) | 10 | 4 | 2 | 7
Erythema infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 6 | 3 | 2 | 6
Gastrointestinal infection (Infections and infestations) | 1 | 1 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 0 | 2 | 1
Influenza (Infections and infestations) | 8 | 2 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4 | 0 | 4
Otitis media (Infections and infestations) | 6 | 3 | 0 | 2
Overgrowth fungal (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 10 | 1 | 2 | 6
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 3
Streptococcal infection (Infections and infestations) | 2 | 5 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 21 | 10 | 2 | 11
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 7 | 1 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 4 | 0 | 2 | 14
Vitamin D decreased (Investigations) | 2 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Joint laxity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1 | 2
Toe walking (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 4 | 2 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 5 | 5 | 2 | 6
Repetitive speech (Nervous system disorders) | 1 | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory processing disorder (Nervous system disorders) | 10 | 5 | 2 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 9 | 7 | 0 | 9
Aggression (Psychiatric disorders) | 22 | 12 | 6 | 14
Agitation (Psychiatric disorders) | 13 | 7 | 6 | 7
Anxiety (Psychiatric disorders) | 1 | 2 | 1 | 2
Apathy (Psychiatric disorders) | 4 | 1 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Defiant behavior (Psychiatric disorders) | 10 | 4 | 4 | 7
Depressed mood (Psychiatric disorders) | 3 | 0 | 1 | 0
Echolalia (Psychiatric disorders) | 3 | 0 | 0 | 1
Encopresis (Psychiatric disorders) | 1 | 0 | 0 | 0
Enuresis (Psychiatric disorders) | 1 | 0 | 0 | 1
Food aversion (Psychiatric disorders) | 1 | 0 | 0 | 0
Frustration tolerance decreased (Psychiatric disorders) | 4 | 2 | 2 | 4
Impulsive behavior (Psychiatric disorders) | 3 | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 11 | 2 | 5 | 6
Intentional self-injury (Psychiatric disorders) | 4 | 3 | 2 | 1
Irritability (Psychiatric disorders) | 6 | 3 | 0 | 3
Negativism (Psychiatric disorders) | 3 | 2 | 1 | 0
Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infection (Psychiatric disorders) | 1 | 0 | 0 | 0
Separation anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Social avoidant behavior (Psychiatric disorders) | 1 | 1 | 0 | 0
Stereotypy (Psychiatric disorders) | 16 | 6 | 1 | 6
Tic (Psychiatric disorders) | 2 | 1 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Aversion (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Gastrointestinal dyskinetic disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 2
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Food refusal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gluten sensitivity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Nipple swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Myringotomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Tooth repair (Surgical and medical procedures) | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02847182/Prot_SAP_000.pdf